CLINICAL TRIAL: NCT06617806
Title: Advanced Practice Nurses for Fall Incidence PrevenTion in Robust Very Old Adults: Protocol for the APN-FIT Hybrid Randomized Controlled Trial
Brief Title: Advanced Practice Nurses for Fall Incidence PrevenTion in Very Old Robust Adults
Acronym: APN-FIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: Pôle Fédératif de Soins Primaires (https://dmg.univ-nantes.fr/c/pole-federatif) (Unknown); UniversitÃ© de Nantes (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RC23_0018; Mécénat AXA 2022 (Other Grant/Funding Number: AXA Life Insurance Company)
Record Dates: First submitted 2024-09-26; First posted 2024-09-27 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Fall Prevention; Autonomy of Older People; Frail Elderly; Advanced Practice Nursing
Keywords: Fall prevention; Aging; Frailty - robustness; Advanced practice nurses; Very old adults

STUDY DESIGN:
Intervention Model Description: Pragmatic randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Advanced Practice Nurse Follow-up (Experimental): The patient is followed-up by his Advanced Practice Nurse and General Practitionner
  The Advanced Practice Nurse (APN) will schedule follow-ups at 1, 3, 6, 9, and 12 months post-inclusion, leveraging their full range of skills and scope of practice. At each follow-up, the APN will ensure that the initial recommendations are being followed and will adjust them according to the patient's progress. The APN will work closely with all actors involved, including the adapted physical activity professional, attending physician, pharmacist, care assistant, and nurse.
  As for all participants, two CGAs will be performed at inclusion by APN and at M12 by the research nurse.
  An Adapted Physical Activity (APA) program will also be included. Participants will receive an APA falls prevention program consisting of 14 sessions, each lasting 45 minutes, conducted by a professional APA teacher in the comfort of their own home.
  Interventions: Other: Follow-up by the Advanced Practice Nurse
- Usual Care (No Intervention): Short version: The patient is handled by his General Practitionner as usual after the first CGA
  Extended version: As for all participants, two CGAs will be performed at inclusion by APN and at M12 by the research nurse.
  An Adapted Physical Activity (APA) program will also be included. Participants will receive an APA falls prevention program consisting of 14 sessions, each lasting 45 minutes, conducted by a professional APA teacher in the comfort of their own home.

INTERVENTIONS:
Other: Follow-up by the Advanced Practice Nurse — At each follow-up (FU), the recommendations of an APN may include :
  * Referral to a specialized memory assessment in case of cognitive impairment
  * Psychological FU in the event that APN detects any mood complaints
  * Ophthalmological and/or ear, nose, and throat consultation if any auditory or visual difficulties is observed
  * Compression stockings use if orthostatic hypotension is present
  * Nutritional counseling, with particular emphasis on the intake of protein, in combination with long-term assessment of weight
  * Supplementation with vitamin D and calcium based to prevent osteoporosis in older adults, especially those at risk of recurrent falls
  * Proposal of a standardized and personalized physical activity program
  * Evaluation of medication therapies, especially antipsychotics, blood pressure medication or broad anticholinergics. The STOPPFall tool will be also proposed and coordinated by APN in accordance with the patient's physician
  * A comprehensive social evaluative approach
  Arms: Advanced Practice Nurse Follow-up

SUMMARY:
APN-FIT is a hybrid type 1 clinical trial comparing the effect of an APN delivered fall prevention programme with standard care in non-frail patients. All participants will receive a full geriatric assessment at enrolment and, on a voluntary basis, physical activity programmes during the 12-month period. Falls occurring during the study will be recorded at 2, 4, 6, 8, 10 and 12 months after enrolment. An ancillary study will specifically examine implementation outcomes of the tested intervention.

DETAILED DESCRIPTION:
Introduction and objectives

The 2020s witnessed the emergence of Advanced Practice Nurses (APN) as a novel paramedical profession in France, bolstering the primary care workforce and service landscape. These nurses are expected to reinforce various dimensions of primary care, including therapeutic education, prevention, screening, and clinical and therapeutic follow-up of patients. There is a need regarding the evaluation of APN led intervention in the prevention of falls in non-frail elderly.

APN-FIT is a pragmatic, hybrid type 1, multicenter, randomized open-label superiority trial addressing this question. The study population will include primary care patients aged over 80 years old, classified as vigorous (according to Clinical Frailty Scale) and able to follow a tailored intervention program. The study will be conducted in seven local primary-care centers in the Pays de la Loire region of France.

Preselection will be done by GPs and APNs, recruitment will be done by APNs in their local caregiving center. APNs will perform a complete comprehensive geriatric assessment (CGA) for each participant at enrolment, followed by a detailed analysis of the resulting data and the emission of a panel of recommendation. A 1:1 randomization of participants will be conducted using a random block size ranging from 4 to 6, stratified by APN.

All participants will benefit from a CGA at inclusion and M12. A home-based physical activity program, over a period of 7 weeks, with twice-weekly sessions (45 min each), will also be proposed to all participants. In the intervention group, each APN will schedule follow-ups at 1, 3, 6, 9, and 12 months post-inclusion. Each participant will be contacted every two months (i.e 2,4,6,8,10 onths) by the research assistant or nurse for data collection on falls and secondary outcome criteria in a blinded approach. All participants will be assessed for a new CGA at M12 by a research nurse.

Quantitative main analysis

The primary outcome is the number of falls recorded at 12 months.

Secondary outcomes include:

* Number of falls and severe falls as defined by the World Fall Guidelines at each time point
* Level of independence, evaluated by Katz' index and Lawton's instrumental activities of daily living
* Level of healthcare utilization
* Level of emergency care service utilization
* Frailty measured with the Clinical Frailty Scale and ICOPE monitor score
* Cognitive performance
* Mental health status
* Nutritional status
* Quality of life evaluated by EQ-5D-5L

A cost-utility analysis (CUA) will be conducted, from a collective perspective and one-year time horizon.

Ancillary study of implementation

An ancillary study will be conducted to facilitate a deeper understanding of the efficacy elements observed in the main study. Its purpose is to determine optimal implementation conditions for practical deployment in the field. The data collection for this ancillary study is primarily opportunistic, coinciding with the data collection necessary to address the main study's primary objective. The indicators described by Proctor and colleagues will be used for the evaluation : acceptability, relevance, adoption, efficiency, feasibility, fidelity, scope and sustainability.

The implementation will undergo evaluation at patient level and healthcare provider level. Individual and group interviews will be conducted. Discourse saturation will be sought. The survey of professionals will occur during initial observations and focus groups. The data analysis will draw from the sociology of professions. A sequential thematic analysis of discourse and a visual examination of non-verbal communication elements and social interactions will be used to capture factors that facilitate or limit program implementation.

ELIGIBILITY:
Inclusion criteria:

* Aged 80 or over;
* Vigorous according to the " Clinical Frailty Scale " (scores 1, 2, 3) ;
* Having a referring primary care physician working in pairs with the local Advanced Practice Nurse;
* affiliated to a Health Care Plan
* Informed and having signed consent to participate in the research.

Exclusion criteria:

* Under guardianship or trusteeship;
* Unable to travel to the primary care office or unable to follow the adapted physical activity program;
* Poor understanding of French.

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 386 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Number of falls in each group | 12 months after enrollment in the study
  An unexpected event in which an individual comes to rest on the ground, floor, or lower level

SECONDARY OUTCOMES:
Number of falls and severe falls at each time point | 2-4-6-8-10 and 12 months after inclusion
  Severe falls is defined by the World Fall Guidelines (2022) as "fall with injuries that are severe enough to require a consultation with a physician; result in the person lying on the ground without capacity to get up for at least one hour; prompt a visit to the emergency room (ER); associated with loss of consciousness"
Level of independance | 12 months after inclusion
  Activities of daily living (Katz index) and Lawton's instrumental activities of daily livng
Level of healthcare utilization | 12 months after inclusion
  Number of consultations, utilization of dental, ophthalmological, and ear-nose-throat care during the follow-up period
Level of emergency care service utilization | 12 months after inclusion
  Number of stays in an emergency hospitalization unit during the follow-up period.
Cognitive performance and mental status | 12 months after inclusion
  MMSE (mini mental state examination) and FAB (frontal assessment battery) score for cognition. Mini-geriatric depression scale for mental health
Quality of Life | 12 months after inclusion
  Evaluated by EQ-5D-5L scale
Frailty and physical performance | 12 months after inclusion
  Frailty measured by the Clinical Frailty scale and Integrated Care for Older People (ICOPE) Monitor score Physical performance assessed with Timed Up and Go test and the Short Physical Performance Battery
Number of participants with malnutrition | 12 months after inclusion
  Body mass index, weight loss and Mini Nutritional Assessment

OTHER OUTCOMES:
Cost utility analysis | 12 months after inclusion
  Rate of Differential Cost - Utility
Implementation outcomes of the intervention | 12 months after the end of the study
  * Acceptability: Perception, among caregivers, that a given treatment, service, practice, or innovation is satisfactory
  * Relevance: Perception of the adequacy of the innovation to address a particular question or problem
  * Adoption: Intention, initial decision, or action to try or use an innovation
  * Efficiency: Assess the price that society is willing to pay to guarantee the health gain associated with the intervention
  * Feasibility: The extent to which an innovation can be successfully implemented within a given organization
  * Fidelity: The degree to which an intervention has been implemented as prescribed in the original protocol
  * Scope: Number of people affected by an intervention and their representativeness of the target population
  * Permanence: The presence of continuity beyond the study regarding the health benefits for the population related to the intervention and the means put in place to ensure it

CONTACTS AND LOCATIONS:
Overall Officials: Laure DE DECKER, MD - Pr, Principal Investigator — Nantes University Hospital
Locations (1):
- CHU Nantes, Nantes, Loire-Atlantique, France

IPD SHARING:
Plan to Share IPD: Yes
A minimal dataset that allows to interpret, replicate and build upon the findings will be available from the corresponding author on reasonable request.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: 12 months after primary publication
Access Criteria: Agreement

REFERENCES:
- [Derived] Huet J, Rat C, Renaux C, Mayol S, Costanza S, Riche VP, Deschamps T, Caillet P, de Decker L. Advanced practice nurses for fall incidence prevention in robust very old adults: protocol for the APN-FIT hybrid randomized controlled trial. BMC Geriatr. 2025 Nov 22;26(1):68. doi: 10.1186/s12877-025-06781-0. PMID 41275104